CLINICAL TRIAL: NCT00047645
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase III Study of the Safety and Efficacy of Subcutaneous Recombinant Interferon-Gamma 1b in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: A Study of the Safety and Efficacy Interferon-Gamma 1b in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: InterMune (Industry)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GIPF-001
Record Dates: First submitted 2002-10-09; First posted 2002-10-11 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2007-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: lung; IPF
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Interferon-gamma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Interferon-gamma 1b — 200 mcg, SQ, 3x per week

SUMMARY:
Study GIPF-001 is phase 3 study designed to determine the safety and efficacy of IFN-g 1b administered by subcutaneous injection; compared to placebo in patients with IPF who are unresponsive to steroids. 330 patients have been enrolled and were assigned to either a IFN-g 1b group or a placebo group.

ELIGIBILITY:
Male or Female, 20-79 years old

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2000-04; Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival time | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Javier Szwarcberg, MD, Study Director — InterMune
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Wells AU, Jacob J, Sverzellati N, Cross G, Barnett J, De Lauretis A, Antoniou K, Weycker D, Atwood M, Kirchgaessler KU, Cottin V. A formula for predicting emphysema extent in combined idiopathic pulmonary fibrosis and emphysema. Respir Res. 2024 Jan 18;25(1):33. doi: 10.1186/s12931-023-02589-x. PMID 38238788
- [Derived] Cottin V, Hansell DM, Sverzellati N, Weycker D, Antoniou KM, Atwood M, Oster G, Kirchgaessler KU, Collard HR, Wells AU. Effect of Emphysema Extent on Serial Lung Function in Patients with Idiopathic Pulmonary Fibrosis. Am J Respir Crit Care Med. 2017 Nov 1;196(9):1162-1171. doi: 10.1164/rccm.201612-2492OC. PMID 28657784